CLINICAL TRIAL: NCT04501445
Title: Relieving the Burden of Psychological Symptoms Among Families of Critically Ill Patients With COVID-19
Brief Title: Psychological Symptoms and Families of COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Central Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20071101
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-07

CONDITIONS: Family Members; Post Intensive Care Unit Syndrome; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rounding Summary (Experimental): Surrogates who were assigned to the intervention group received a written rounding summary every day or every other day that the patient is in the ICU.
  Interventions: Behavioral: Written Summary of Rounds
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Written Summary of Rounds — The summary was organized as follows for each of the most important ICU problems: 1) Description of the problem, 2) Ways the ICU team is addressing the problem i.e. consultations, diagnostic tests, and treatments. 3) An assessment of whether the problem is improving or worsening.
  Arms: Rounding Summary

SUMMARY:
Families of patients in Intensive Care Units (ICUs) are at increased risk for developing psychological symptoms that can last for months after the patient is discharged. These symptoms can have significant impact on both the patient and family member's quality of life.

The investigators have found that families of patients admitted to the Rush University Medical Center ICU during to the COVID-19 pandemic were more likely to develop clinically significant psychological symptoms than families of patients admitted prior to the COVID-19 pandemic. The investigators suspect that this finding is due in part to the hospital-wide no visitation policy that altered our standard communication practices and may have prevented families from being active participants in the patient's medical care.

The goals of this project are 1) to determine the prevalence of psychological disorders among families of COVID-19 patients after ICU discharge 2) to determine the characteristics of ICU care that were associated with the development of psychological disorders among family members and 3) to pilot a program in which families with psychological disorders after ICU discharge receive therapy from mental health professionals.

DETAILED DESCRIPTION:
Part 1- Post-ICU discharge survey and Interview Upon enrollment in this post-ICU discharge follow-up study, the subject (surrogate of the ICU patient) will complete a survey dealing with the patient's course since Rush discharge

1. Is the patient still alive?

   1. If deceased, did the patient pass away at Rush or after discharge from Rush?
   2. If alive, is the patient at home?

   i. If at home, for how long? Is he/she receiving home health services?
2. If the patient did not pass away at Rush, did the patient spend time in a rehabilitation hospital, nursing home, or long-term acute care hospital after discharge from Rush?
3. Is the patient currently having any of the following symptoms (check all that apply).

   1. Fatigue
   2. Trouble Breathing
   3. Difficulty speaking
   4. Difficulty eating
   5. Difficulty thinking or paying attention
   6. Pain or discomfort
   7. Anxiety
   8. Depressed mood
   9. Difficulty moving or walking
   10. Difficulty performing activities of daily living such as dressing or bathing
4. Have the subject used mental health services since the time the patient was admitted?
5. What is the subject's overall impression of mental health services (choices ranging from very unhelpful to very helpful)

Subjects will be asked to complete the 1) Critical Care Family Needs Inventory (CCFNI) questionnaire, 2) Hospital Anxiety and Depression Scale (HADS), and 3) Impact of Events Scale Revised (IES-R) questionnaire.

Subjects will participate in a 30-minute phone interview with a member of the study team. The interviewer will review the subject's responses to the above surveys and ask follow-up questions. The interviewer will ask how the subject has been coping with any psychological symptoms (i.e. anxiety, depression, post-traumatic stress)

The psychologist will describe different types of interventions for people coping psychological symptoms and assess the subject's interest in pursuing any of them.

Part 2 - Post-ICU psychological intervention Subjects with clinically significant psychologist symptoms based on either their survey or interview responses will be invited to participate in 6-week trauma-focused intervention with a psychologist.

The program will be brief and delivered online to test the acceptability and feasible of the program, and to gather a preliminary estimate of effect size. We will pilot a group-based intervention (n =3-5) online over Zoom and deliver the intervention across six sessions outlined below. Sessions will last 60-75 minutes depending on participant questions and discussion. Experiential exercises will be drawn from Acceptance and Commitment Therapy, a related contemporary cognitive behavioral treatment (Hayes, Strosahl, & Wilson, 2012). Some commentary of Viktor Frankl's (1985) work on meaning making will be made in group discussion. Activity scheduling worksheets from Martell, Dimijian and Herman-Dunn (2013) will be used for out of session homework.

We plan two phases for the study. The first phase, sessions 1-3, focus on introducing the model of behavioral activation and guide the participants to identify activities that will being pleasant, meaningful, or offer a sense of accomplishment and mastery. The first session aims to normalize diverse responses to health-related stress and loss by introducing the behavioral model of depression, and the rationale for behavioral activation. In the second session participants then clarify their values, so that they can begin scheduling pleasant and/or meaningful activities in the third session. These activities are tailored based on each participant's individuals goals, priorities and values. The second phase, sessions 4-6, aims to reinforce and sustain positive gains made via behavioral activation and pleasant activity scheduling. Session 4 offers suggestions for problem-solving ways to overcome unhelpful avoidance, a transdiagnostic vulnerability that sustains a number of emotional and psychiatric disorders. Session 5 offers suggestions for overcoming rumination including instruction in mindfulness, and attentional techniques that help participants attend to the outcomes and experiences of the pleasant activities they engage in. Session 6 concludes the program, and guides participants to consider plans to maintain commitment to pleasant activities.

Session 1 Psychoeducation Introductions. Question to group: Why are we here?

* Normalize the grieving process and the challenges of COVID safety guidelines

  * grief, boredom, loneliness
  * 1/3 of USA adults report depression and anxiety
* Discuss the behavioral model of depression - loss of reward and meaningful events as a prelude to negative moods of all types
* Behavioral Activation as a strategy to enhance reward and meaning
* Experiential: Contemplate a time in life when you felt you were doing well. How were you engaging the world around you?
* Homework: Start Activity tracking. Worksheets will be provided, but we allow a more feasible approach of jotting down 1-2 words about activity and providing a subjective mood rating.

Session 2 Value Clarification Question to the group: How do we bring purpose into our living?

* Consider values as the foundation of meaning and purpose
* Discuss meaning in life and Dr. Viktor Frankl's thesis that humans are driven to find meaning

  o "We do not ask life what the meaning of life is. Life asks us, what is the meaning of your life. And life demands our answer."
* What gives/gave meaning to your loved one's life? What would make them smile? If you share values with this person, how can you honor those values you share in your own commitments and activities?
* Experiential: Contemplate your 80th Birthday, Retirement Speech, family remembering you far in the future, etc, Homework: Values Compass. Participants will complete the values compass worksheet in which they rate their perceived importance and engagement in various domains of living (e.g, family life, learning, spirituality).

Session 3 Scheduling Activities Question to group: What does it mean to be committed?

* Discuss a role model or mentor who demonstrated commitment to something important. How did they do it? Do they share values with the patient they care(d) for? How do these
* Selecting and scheduling pleasant events. Regardless of how you feel, take action to experience:

  * Pleasure
  * Mastery
  * Purpose
  * Health habits: steady sleep, diet, exercise
* Experiential: Participants visualize, write or discuss steps needed to engage a plan. Visualize yourself overcoming a roadblock or barrier.
* Homework: Activity Schedule. Participants will schedule several pleasant/meaningful events for the coming week. They will rate their mood while engaged in these activities and journal about their experiences.

Session 4 Overcoming Avoidance What do we do with fear?

* Getting out of the TRAP (Trigger-Response-Avoidance Pattern) to get on Track (Trigger Response Adaptive Coping)
* Often we hurt when something that matters is threatened. We should protect what matters not the momentary feeling. Discuss "fear as an arrow" that can be useful for pointing to ones values (e.g., we typically do not fear losing things we do not care about).
* Experiential: Flipping the coins of avoidance. Participants look to how fears, and frustrations relate to other prosocial and personally valued events and experiences.
* Homework: Activity Schedule. This repeats the homework from the prior week.

Session 5 Working with thoughts Question to the group: How do we prevent going on autopilot so we stay focused on what matters?

* Staying present to notice when actions are working. Being better at tracking outcomes.
* Mindfulness versus rumination
* Experiential: Mindfulness of the present. Participants are guided in a mindfulness exercise to attend to sense experiences in the present moment. The goal of the exercise is to introduce a skill for re-orienting to the present moment. This is particularly needed for attending to and noticing the pleasant and meaningful experiences that come from behavioral activation.
* Homework: Activity Schedule Session 6 Recap and review Question to the group: How do we carry these lessons with us? How do we share these lessons with others?
* The goal of this session is to review and to provide additional practice with any of the prior skills discussed in previous sessions.
* Relapse prevention concepts will be discussed. Participants will be encouraged to continue to maintain pleasant activity scheduling, and to consider how these activities can be reinforced through social commitments, and daily reflection.
* Consider making a symbol. Picture, photo, card, note to self to remind oneself of a valued activity. This can be displayed in a prominent place (e.g., family photo on the mantle, photo of exercise on bathroom mirror, religious text on coffee table). Should evoke pleasant memory, and motivation.

Prior to beginning the intervention and at the completion of the intervention, surrogates will complete the 1) Hospital Anxiety and Depression Scale (HADS), and 2) Impact of Events Scale Revised (IES-R) questionnaire.

At the completion of the intervention, subjects will participate in another 30-minute phone interview with a study investigator. The study investigator will review the subject's responses to the above surveys and ask follow-up questions. The study investigator will ask how the subject has been coping with any psychological symptoms (i.e. anxiety, depression, post-traumatic stress).

All interviews will be audio recorded and transcribed. Two members study staff will review the transcriptions and use thematic content analysis to determine the types of psychological symptoms that are present and the reason(s) they may be present.

When analyzing subject responses, the investigators will account for the following variables

* Whether the patient is deceased or not
* Length of time since hospital discharge
* Whether the subject received mental health services on their own or not
* Whether the subject received daily written summaries in the ICU or not

Statistical Analysis The investigators expect ~100 subjects to meet inclusion criteria. The investigators expect ~70-100 to complete Part 1 (Post-ICU discharge survey and Interview). The investigators will determine the prevalence of psychological symptoms and opinions on ICU care by reviewing survey responses and interview recordings. The investigators expect ~30 to complete Part 2 (Post-ICU discharge survey and Interview). The investigators compare pre- to post-intervention survey responses for each subject using a paired t-test. Part 2 will be considered a pilot study. The investigators will use the results to plan a future, adequately powered study.

ELIGIBILITY:
Inclusion Criteria:

* The patient's surrogate was enrolled in "ICU Rounding Summaries for Families of Critically Ill Patients" (NCT03969810) and the patient had COVID-19
* The patient has been discharged from the hospital

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davidson JE, Jones C, Bienvenu OJ. Family response to critical illness: postintensive care syndrome-family. Crit Care Med. 2012 Feb;40(2):618-24. doi: 10.1097/CCM.0b013e318236ebf9. PMID 22080636
- [Background] Nelson JE, Hanson LC, Keller KL, Carson SS, Cox CE, Tulsky JA, White DB, Chai EJ, Weiss SP, Danis M. The Voice of Surrogate Decision-Makers. Family Responses to Prognostic Information in Chronic Critical Illness. Am J Respir Crit Care Med. 2017 Oct 1;196(7):864-872. doi: 10.1164/rccm.201701-0201OC. PMID 28387538
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Derived] White KR, Lee JJ, Sarigiannis KA, Tringali JJ, Vu J, Eaton England A, Lietzau S, Hebert C, Banayan D, Basapur S, Glover CM, Shah RC, Gerhart J, Greenberg JA. Restrictive Visitation Policies and Related Post-Traumatic Stress Among Families of Critically Ill Patients With COVID-19. Chest. 2023 Dec;164(6):1462-1465. doi: 10.1016/j.chest.2023.06.021. Epub 2023 Jun 24. No abstract available. PMID 37356707
- [Derived] Sarigiannis KA, Tringali JJ, Vu J, Eaton England A, Lietzau S, Hebert C, Banayan D, Basapur S, Glover CM, Shah RC, Gerhart J, Greenberg JA. Symptoms of Anxiety, Depression, and Stress among Families of Critically Ill Patients with COVID-19: A Longitudinal Clinical Trial. Ann Am Thorac Soc. 2023 May;20(5):705-712. doi: 10.1513/AnnalsATS.202209-797OC. PMID 36603135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who completed surveys after ICU discharge
Groups:
- Surveyed After ICU Discharge: Surveyed after ICU discharge
Period: Overall Study
Arm/Group | Surveyed After ICU Discharge
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surveyed After ICU Discharge
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 84
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 14
  More than one race | 0
  Unknown or Not Reported | 58
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Post-Traumatic Stress Disorder (PTSD) Initial
Description: Score on Impact of Events Scale Revised (IES-R) questionnaire. 22 questions. Score 0-88 with higher scores indicating more stress.
Time Frame: Measured once upon enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Surveyed After ICU Discharge: Survey after ICU discharge
Arm/Group | Surveyed After ICU Discharge
Number analyzed (Participants) | 90
score on a scale | 27.9 (17.9)

2. Primary Outcome: Symptoms of Anxiety and Depression Initial
Description: Score on Hospital Anxiety and Depression Scale (HADS). Total score 0-21 for anxiety (7 questions) and 0-21 for depression (7 questions). Higher scores indicate greater symptom burden.
Time Frame: Measured once upon enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveyed After ICU Discharge
Number analyzed (Participants) | 90
score on a scale | 12.8 (8.9)

3. Secondary Outcome: Surrogate Satisfaction With the Patient's ICU Care:
Description: Score on the Critical Care Family Needs Inventory (CCFNI) questionnaire. 14 questions. Total score range 14-56 with lower scores indicating better satisfaction.
Time Frame: Measured once upon enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveyed After ICU Discharge
Number analyzed (Participants) | 90
score on a scale | 16.8 (6.0)

4. Secondary Outcome: Symptoms of Post-Traumatic Stress Disorder (PTSD) Final
Description: IES-R score before intervention
  The IES-R yields a total score (ranging from 0 to 88) with higher scores indicative of more severe PTSD
Time Frame: Measured before behavioral intervention (6-12 weeks after enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Received Group Intervention: Received group intervention
Arm/Group | Received Group Intervention
Number analyzed (Participants) | 26
score on a scale | 36.9 (17.0)

5. Secondary Outcome: Symptoms of Post-Traumatic Stress Disorder (PTSD) Final
Description: IES-R after intervention
  The IES-R yields a total score (ranging from 0 to 88) with higher scores indicative of more severe PTSD
Time Frame: Measured after behavioral intervention (12-24 weeks after enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveyed After ICU Discharge
Number analyzed (Participants) | 19
score on a scale | 24.1 (13.5)

6. Secondary Outcome: Symptoms of Anxiety and Depression Final
Description: as for outcome 2
Time Frame: Measured before behavioral intervention (6-12 weeks after enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveyed After ICU Discharge
Number analyzed (Participants) | 26
score on a scale | 15.9 (9.4)

7. Secondary Outcome: Symptoms of Anxiety and Depression Final
Description: as for outcome 2
Time Frame: Measured after behavioral intervention (12-24 weeks after enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Surveyed After ICU Discharge
Number analyzed (Participants) | 19
score on a scale | 11.7 (7.0)

8. Secondary Outcome: Interview Initial
Description: Qualitative analysis of phone interview to determine the presence and reason(s) for psychological symptoms
Time Frame: Measured once upon enrollment
Reporting Status: Not Posted

9. Secondary Outcome: Interview Final
Description: Qualitative analysis of phone interview to determine the presence and reason(s) for psychological symptoms
Time Frame: Measured after behavioral intervention (12-24 weeks after enrollment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3-6 months after enrollment
Arm/Group | Received Group Intervention
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
small sample size, single center

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT04501445/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04501445/ICF_001.pdf